CLINICAL TRIAL: NCT00002398
Title: A Randomized, Open-Label Expanded Access Program to Evaluate the Safety of Preveon (Adefovir Dipivoxil) at Two Dose Levels When Used in Combination With Other Antiretroviral Agents for the Treatment of Patients With HIV Infection Who Have Failed Other Antiretroviral Therapy and Have Limited Treatment Options
Brief Title: Safety and Effectiveness of Giving Adefovir (Preveon) Plus Other Anti-HIV Drugs to HIV-Infected Patients Who Have Not Responded to Other Anti-HIV Drug Combinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 232G; GS-97-423
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-12

CONDITIONS: HIV Infections
Keywords: HIV-1; Acquired Immunodeficiency Syndrome; Adenine; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Carnitine; adefovir dipivoxil

INTERVENTIONS:
Drug: Levocarnitine
Drug: Adefovir dipivoxil

SUMMARY:
The purpose of this study is to see if it is safe and effective to give adefovir plus other anti-HIV drugs to HIV-infected patients who have failed other anti-HIV drug combinations. This study will try to make adefovir available to all AIDS patients who need it.

Some patients do not respond to anti-HIV drug combinations, even when different combinations are tried. Adefovir may be able to help these patients fight HIV.

DETAILED DESCRIPTION:
Recent studies indicate that the use of triple-combination therapy, in particular the combinations of reverse transcriptase inhibitors and a protease inhibitor, can result in a significant decrease in plasma HIV-1 RNA levels and an increase in CD4 cell count. Continued follow-up of patients taking triple-combination drug regimens has in some cases demonstrated sustained suppression of plasma HIV-1 RNA levels for up to 18 months. Furthermore, despite the potent antiviral effect of some triple combinations, a percentage of patients continue to have measurable levels (more than 500 copies/ml) of HIV-1 RNA in plasma, even when treated with a combination of 2 reverse transcriptase inhibitors and indinavir. Over time, some patients experience a rebound of plasma HIV-1 RNA for reasons that are not well understood. [AS PER AMENDMENT 7/8/98: Randomization to 2 dose levels may allow more patients to derive therapeutic benefit from Preveon by minimizing adverse effects.]

Patients not previously enrolled in clinical trials of Preveon are randomized to 1 of 2 doses of Preveon orally once daily and L-carnitine orally once daily. [AS PER AMENDMENT 7/8/98: Patients must receive other antiretroviral agents concomitantly with Preveon; at least 1 other antiretroviral agent must be added with Preveon that was not previously administered to the patient.Patients previously enrolled in Preveon clinical trials who "roll in" to expanded access and who have received at least 16 weeks of Preveon receive open-label Preveon orally once daily and L-carnitine orally once daily, taken with or without food at the same time each day.] All patients enrolled in expanded access are randomized in a 1:1 fashion to 1 of 2 doses taken orally once daily. Patients initially assigned to the higher dose will have their Preveon dose reduced to the lower dose at Week 16 of treatment. Patients initially assigned to the lower dose continue this dose unless dose modification to an even lower dose for toxicity is required. [AS PER AMENDMENT 7/8/98: Additional informed consent is needed for this reduction due to limited efficacy of the lower dosage in treating HIV infection.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 cell count of 50 cells/mm3 or less within the past 2 months.
* Have a viral load (level of HIV in the body) of 30,000 copies/ml or more within the past 2 months.
* Are at least 13 years old (need consent of parent or guardian if under 18).
* Have failed to respond to an anti-HIV drug combination that included at least 2 nucleoside reverse transcriptase inhibitors and at least 1 protease inhibitor (PI).
* Do not have any other anti-HIV treatment options left.
* Agree to use effective methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have certain serious medical conditions that would prevent you from completing the study, including serious kidney disorders.
* Have taken certain medications, including certain treatments for opportunistic (HIV-related) diseases.
* Are pregnant or breast-feeding.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Gilead Sciences Inc, Foster City, California, United States